CLINICAL TRIAL: NCT04823572
Title: Efficacy of a New-generation Platelet-Rich Fibrin in the Treatment of Periodontal Intrabony Defects : a Randomized Clinical Trial
Brief Title: Treatment of Periodontal Intrabony Defects With A-PRF or OFD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SE TUKEB 254/2017
Record Dates: First submitted 2021-03-04; First posted 2021-04-01 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2022-04

CONDITIONS: Periodontal Diseases
Keywords: Intrabony Defects; Periodontal Regeneration; A-PRF; Advanced Platelet-Rich Fibrin; Open Flap Debridement
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-PRF Advanced Platelet-Rich Fibrin (Active Comparator): Comparing healing effect of an autologous product with open flap debridement.
  Interventions: Procedure: A-PRF/OFD
- OFD Open Flap Debridement (Active Comparator): Comparing healing effect of an autologous product with open flap debridement.
  Interventions: Procedure: A-PRF/OFD

INTERVENTIONS:
Procedure: A-PRF/OFD — Comparing healing effect of an autologous and open flap debridement

SUMMARY:
The aim of this randomized clinical trial was to clinically evaluate and compare the healing of intrabony defects after treatment with advanced platelet-rich fibrin (A-PRF+) toped flap debridement (OFD) in periodontitis patients.

DETAILED DESCRIPTION:
Thirty (30) intrabony defects are randomly divided in two treatment groups: test (n = 15) and control (n = 15). The intrabony defects are filled with A-PRF+ (n=15) in the test group, respectively treated with open flap debridement in the control group, and fixed with sutures to ensure wound closure and stability.

ELIGIBILITY:
Inclusion Criteria:

* no systemic diseases
* a good level of oral hygiene
* presence of a 2-, 3-, or combined 2-3-wall intrabony defect with a defect angle of 20-40 (+/- 5) degrees
* with a minimum PPD of 6 mm and intrabony component of a minimum 4 mm as detected on radiographs
* no smoking

Exclusion Criteria:

* systemic diseases that could influence the outcome of the therapy
* poor oral hygiene
* smoking
* horizontal bone loss

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Periodontal clinical parameters | Change from baseline after 6 month and after 12 month
  to determine the clinical attachment level (CAL) With a calibrated periodontal probe we are examining the changes of periodontal probing depth (PPD) and gingival recession (GR) after surgical procedure in mm, the two parameters are used to determine the clinical attachment level (CAL).

CONTACTS AND LOCATIONS:
Overall Officials: Dőri Ferenc, Professor, Principal Investigator — Semmelweis University
Locations (1):
- Semmelweis University, Department of Periodontology, Budapest, Hungary